CLINICAL TRIAL: NCT04899622
Title: Mindfulness Combined With Virtual Exercise Online (MOVE) Compared With a Self-Management Guide for Adults With Chronic Pain: Study Protocol for a Feasibility Randomised Controlled Trial
Brief Title: Mindfulness Online and Virtual Exercise (MOVE) Compared With Self-Management for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orla Deegan (Other)
Collaborators: Mater Misericordiae University Hospital (Other); University College Dublin (Other)
Responsible Party: Sponsor-Investigator, Orla Deegan, Prinicipal Investigator, University College Dublin
Organization: University College Dublin (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOVE-Online
Record Dates: First submitted 2021-04-20; First posted 2021-05-24 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Pain Management Programme; e-Health; Mindfulness Based Stress Reduction; Exercise
MeSH Terms: conditions — Chronic Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined MBSR and exercise (Experimental): Group A will take part in live online weekly mindfulness sessions based on the Mindfulness Based Stress Reduction (MBSR) programme, in addition to supervised exercise classes.
  Interventions: Behavioral: MBSR; Behavioral: Exercise
- Online Self-Management Guide (Active Comparator): Group B will be invited to interact with an online self-management guide accessible in the members area of the study website.
  Interventions: Behavioral: Online Self-Management Guide

INTERVENTIONS:
Behavioral: MBSR — Participants will attend weekly online classes (two hours duration) of MBSR for eight weeks. The classes will be delivered live online to groups of up to fifteen participants and will be led by Mindfulness instructors with MSc degrees in Mindfulness Based Interventions. The programme content will be based on the standard MBSR programme and is tailored towards key concerns and difficulties experienced by individuals with chronic pain.
  Arms: Combined MBSR and exercise
Behavioral: Exercise — Participants will attend weekly classes of supervised classes (1 hour) for eight weeks, following the MBSR class. The exercise class will be delivered live online to the group by an experienced Physiotherapist and will consist of a range of flexibility and strengthening exercises which will be advanced every two weeks for the duration of the eight week programme. The exercises will also be available in video format on the mobile application "Physitrack" which each participant will be invited to download. This will allow the participants to review the exercises between sessions, record online if they have completed each exercise and in addition rate their pain experience while completing the exercises.
  Arms: Combined MBSR and exercise
Behavioral: Online Self-Management Guide — Participants will receive standard evidence based self-guided information which they will access independently via the members area of the study website. This 'Online Self-Management Guide' will consist of eight categories of self-management; (1) What is chronic pain? (2) Chronic pain and nutrition (3) Sleep issues with chronic pain (4) Activity and exercise (5) Pacing (6) Using a pain diary (7) Relaxation and mindfulness and (8) Course summary. The information will be presented in the form of general text, links to online resources and videos. The information in this area will be updated biweekly during the eight week programme with the participants receiving bi-weekly email reminders.
  Arms: Online Self-Management Guide

SUMMARY:
The aim of this study is to assess the feasibility and acceptability of a combined Mindfulness Based Stress Reduction (MBSR) and exercise online programme compared to an online self-management guide. Pain management programmes are the recommended treatment for chronic pain, however a number of barriers to their widespread implementation have been identified including geographical distance from speciality programmes, functional disability limiting the mobility of people with CP and economic limitations(1). eHealth interventions have the potential to address a number of these barriers and recent reviews have reported reductions in pain(2), improved knowledge and understanding about chronic pain and chronic pain management, improved function(3) and improvements in quality of life(4) following eHealth interventions.

The intervention in this study will be delivered online. Participants will be randomly allocated to a combined MBSR and exercise programme (Group A) or an online self-management guide (Group B). Group A will take part in an 8 week live online weekly mindfulness sessions based on the Mindfulness Based Stress Reduction (MBSR) programme facilitated by a qualified mindfulness teacher, in addition to a supervised exercise classes led by a Physiotherapist. Group B will receive access to an 8 week online self-management guide containing 8 self-directed guides, which will be made available to participants biweekly.

Outcomes of feasibility and acceptability will be investigated in addition to a preliminary examination of between group clinical effects at baseline immediately post intervention and at a three month follow up, using validated patient reported outcome measures. In addition all participants will wear a Fitbit activity monitor for the duration of the eight-week interventions to capture activity measures. A qualitative study will also be conducted to gather participants' perceptions of the programme and its usefulness

DETAILED DESCRIPTION:
This study is a parallel-groups, randomised-controlled, feasibility trial. Seventy-five participants aged 18 years and over, who have been diagnosed with a chronic pain condition by a Consultant in Pain Medicine or a General Practitioner will be recruited to the feasibility study. Participants will be individually randomised to one of two interventions. Group A will take part in live online weekly mindfulness sessions based on the Mindfulness Based Stress Reduction (MBSR) programme facilitated by a qualified mindfulness teacher, in addition to supervised exercise classes led by a Physiotherapist. The combined 3 hour intervention (2 hours MBSR, 1 hour exercise) will take place one day per week for 8 weeks. Group B will receive access to an 8 week online self-management guide containing 8 self-directed guides, with the material released biweekly.

The key outcomes measures will include; (1) recruitment rates, eligibility rates, willingness to be randomised; (2) feasibility and acceptability of data collection instruments and procedures; (3) intervention adherence, engagement and attrition rates; (4) feasibility and acceptability of the interventions and; (5) participants' subjective perceptions of the programmes.

The study will also include a preliminary examination of between group clinical effects at baseline, immediately post intervention and at a three month follow up, using the following validated patient reported outcome measures; Pain Self-Efficacy Questionnaire, Brief Pain Inventory, Pain Catastrophizing Scale, Generalised Anxiety Depression Assessment, Patient Health Questionnaire-9, Pain Disability Index, Fear Avoidance Belief Questionnaire, Short-Form-36 Health Survey, Patient Global Impression of Change Scale and measure of treatment satisfaction adapted from the Client Satisfaction Questionnaire (CSQ-8).

Physical activity levels (average daily step count, distance travelled and active minutes) will be measured for all participants using Fitbit Charge 4 activity monitors for the duration of the eight-week intervention period.

Analyses of the feasibility study will primarily be descriptive and will address the outcomes relating to the feasibility and acceptability of the interventions and the procedures of the study. Between-group comparisons of clinical treatment effects will be descriptive and exploratory to consider the viability of the combined MBSR and exercise intervention that may warrant further exploration in a fully powered RCT.

A sample of participants will be invited to attend focus groups where semi-structured interviews will be conducted with the aim of gathering information on the participants' subjective perceptions of the programme and its usefulness.

ELIGIBILITY:
Inclusion criteria:

•. Aged >18 years

* Diagnosis of chronic pain by a Consultant in Pain Medicine or General Practitioner
* Presence of pain NRS ≥ 3 of greater than three months' duration
* Ability to provide informed consent
* Ability to communicate in English and understand English

Exclusion criteria:

* Need for further diagnostic evaluation (determined by doctor)
* Presence of any contraindications to participation in an exercise programme E.g. severe shortness of breath at rest, angina, uncontrolled diabetes or epilepsy, recent (previous 3 weeks) myocardial infarction, pulmonary embolism, deep vein thrombosis or asthma attack.
* Presence of active cancer
* Concurrent participation (or in the previous 3 months) with any form of psychological, physiotherapy or supervised exercise in addition to the study intervention.
* Presence of substance misuse (diagnosed by the Pain Consultant/GP).
* Inability to take part in an online exercise programme
* Standard MBSR exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Number of eligible participants identified per programme | Baseline
  Prior to each programme the number of eligible participants will be recorded by the primary researcher
Number of eligible participants recruited per programme | Baseline
  Prior to each programme the number of eligible participants who are recruited will be recorded by the primary researcher
Reasons for non-participation | Baseline
  This measure will be recorded by the primary researcher when screening participants
Number of participants who complete the study | immediately post intervention (8 weeks from baseline)
  The number of participants that complete >50% of the online classes programme
Adherence to completion of baseline patient reported outcome measures | Baseline
  Numbers of participants completing > 90% of baseline patient reported outcome measures
Adherence to completion of immediate follow-up patient reported outcome measures | Immediately post intervention (8 weeks from baseline)
  Numbers of participants completing > 90% of follow-up patient reported outcome measures
Adherence to completion of long term follow-up patient reported outcome measures | 3 months post intervention (20 weeks from baseline)
  Numbers of participants completing > 90% of follow-up patient reported outcome measures
Interaction with online self-management guide | Immediately post intervention (8 weeks from baseline)
  The study website analytics will measure the number of views that each element of the online guide receives (Group B)
Treatment Acceptability (Satisfaction assessed by Client Satisfaction Questionnaire-8) | Immediately post intervention (8 weeks from baseline)
  Patient satisfaction with treatment will be measured with an adapted version of the Client Satisfaction Questionnaire-8. Responses are scored from 1-4, and the possible total scores range from 8 to 32. Higher scores indicate greater satisfaction.
Interface usability | immediately post intervention (8 weeks from baseline)
  Measures of website usability will be investigated with an adapted System Usability Scale (SUS) Scores range from 10-50. Higher scores indicated greater ease of usability.

SECONDARY OUTCOMES:
Change in pain self-efficacy measured with the Pain Self-Efficacy Questionnaire | immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  The Pain Self-Efficacy Questionnaire is a ten item questionnaire which assesses an individual's confidence in their ability to perform a variety of activities or tasks despite pain. Scores can range from 0 - 60. Higher scores represent lower confidence to function with pain.
Change in symptoms of anxiety measured with the Generalized Anxiety Disorder Assessment | immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  The Generalized Anxiety Disorder 7 assesses symptoms of anxiety experienced during the last two weeks. The total score for the seven items ranges from 0 to 21. Higher scores represent higher levels of anxiety.
Changes in symptoms of depression measured with the Patient Health Questionnaire 9 | immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  Symptoms of depression will be assessed using the Patient Health Questionnaire 9, which is a nine-item questionnaire generating scores ranging from 0-27. Higher scores indicate increased severity of depression.
Changes in pain severity and pain interference measured with the Brief Pain Inventory-Composite pain score | immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  Pain severity will be measured using the pain severity subscale of the Brief Pain Inventory. Pain interference will be measured using the interference subscale of the Brief Pain Inventory, which measures the extent to which pain interferes with functions such as general activity, walking ability, normal work, mood, relationships with people, enjoyment of life and sleep. For each scale, the total score is the average of all items (range, 0-10), where a higher score indicates greater severity and more interference.
Changes in the impact of pain on individuals life participation measured with the Pain Disability Index | immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  The Pain Disability Index measure asks patients to rate how much pain interferes in seven areas of life activity: family/home, recreation, social, occupation, sexual, self-care and life-support. Total score ranges from 0-70. The higher the score the greater the person's disability due to pain.
Changes in fear avoidance of physical activity measured with the Fear Avoidance Belief Questionnaire. | immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  The Fear Avoidance Belief Questionnaire measures patients' fear of pain and consequent avoidance of physical activity because of their fear. The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. The scores range from 0-96; higher scores indicates increased fear avoidance behaviours.
Change in pain catastrophising measured with the Pain Catastrophising Scale. | immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  The Pain Catastrophising Scale is a 13-item instrument designed to assess catastrophic thinking in relation to pain. It yields a total score and three subscale scores assessing rumination, magnification and helplessness. Scores range from 0-52. Higher scores are associated with higher amounts of pain catastrophising.
Change in quality of life measured with the Short Form-36 Health Survey | immediately post intervention (8 weeks from baseline) and 12 week follow up (20 weeks from baseline)
  The Short Form-36 Health Survey comprises of 36 questions which cover eight domains of general health. Scores range from 0-100. The lower the score the more disability.
Patient Global Impression of Change Scale | immediately post intervention (8 weeks from baseline)
  The Patient Global Impression of Change Scale scale measures a patient's rating of overall improvement or lack thereof due to the intervention. It is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Changes in step count (Fitbit) | immediately post intervention (8 weeks from baseline)
  Average weekly step count will be measured using a Fitbit Charge 4 activity monitor worn by participants for the eight weeks of the intervention.
Changes in distance travelled (Fitbit) | immediately post intervention (8 weeks from baseline)
  Average weekly distance travelled will be measured using a Fitbit Charge 4 activity monitor worn by participants for the eight weeks of the intervention.
Changes in active minutes (Fitbit) | immediately post intervention (8 weeks from baseline)
  Average active minutes will be measured using a Fitbit Charge 4 activity monitor worn by participants for the eight weeks of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Doody, Study Director — University College Dublin
Locations (1):
- University College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keogh E, Rosser BA, Eccleston C. e-Health and chronic pain management: current status and developments. Pain. 2010 Oct;151(1):18-21. doi: 10.1016/j.pain.2010.07.014. Epub 2010 Jul 31. No abstract available. PMID 20674174
- [Background] Macea DD, Gajos K, Daglia Calil YA, Fregni F. The efficacy of Web-based cognitive behavioral interventions for chronic pain: a systematic review and meta-analysis. J Pain. 2010 Oct;11(10):917-29. doi: 10.1016/j.jpain.2010.06.005. Epub 2010 Jul 22. PMID 20650691
- [Background] Bender JL, Radhakrishnan A, Diorio C, Englesakis M, Jadad AR. Can pain be managed through the Internet? A systematic review of randomized controlled trials. Pain. 2011 Aug;152(8):1740-1750. doi: 10.1016/j.pain.2011.02.012. Epub 2011 May 11. PMID 21565446
- [Background] Mariano TY, Wan L, Edwards RR, Jamison RN. Online teletherapy for chronic pain: A systematic review. J Telemed Telecare. 2021 May;27(4):195-208. doi: 10.1177/1357633X19871746. Epub 2019 Sep 5. PMID 31488004
- [Derived] Deegan O, Fullen BM, Casey MB, Segurado R, Hearty C, Doody CM. Combined online interactive mindfulness and exercise programme (MOVE-Online) compared with a self-management guide for adults with chronic pain: protocol for a randomised controlled feasibility trial. BMJ Open. 2022 Feb 9;12(2):e058265. doi: 10.1136/bmjopen-2021-058265. PMID 35140163